CLINICAL TRIAL: NCT06774586
Title: Study of the Characteristics of the Vascular Wall in Pediatric Age
Acronym: PEDVASC
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PEDVASC
Record Dates: First submitted 2024-12-01; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-10

CONDITIONS: Cardiovascular Diseases
Keywords: vascular wall; pediatrics
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With this study, we want to investigate the characteristics of the blood vessel wall and study cardiovascular risk in children and adolescents, whether or not they have heart disease, by subjecting patient to a noninvasive diagnostic examination with an innovative medical device called VICORDER©.

DETAILED DESCRIPTION:
Cardiovascular (CV) disease remains the leading cause of death in adulthood in industrialized countries, and processes of vascular wall disruption are a key pathogenetic element of this. These processes can begin as early as childhood, contributing to CV risk in later ages.

In particular, increased arterial stiffness is an independent CV risk factor that is associated with increased mortality, and its measurement may influence therapeutic decisions. The clinical value of studying arterial stiffness is recognized by the European Network for Noninvasive Investigation of Large Arteries and the 2018 European Society of Cardiology guidelines on hypertension.

The method considered as the gold standard for measuring arterial stiffness is carotid-femoral Pulse Wave Velocity (PWV), which can be measured noninvasively. The stiffer the arterial wall, the more PWV increases; left ventricular afterload and systolic arterial pressure (SAP) increase, while diastolic arterial pressure (DAP) and coronary perfusion decrease. Increased afterload promotes left ventricular hypertrophy, with increased oxygen demands, and thus increased susceptibility to myocardial ischemia.In pediatric age, the most important CV risk factors include overweight and obesity, hypertension (which, between 0 and 18 years has a prevalence of 3-5%, alterations in glucose and lipid metabolism, diabetes mellitus, and kidney disease, especially chronic renal failure. These risk factors promote increased arterial stiffness and thus the risk of adverse events.Some typical pediatric vasculitides can also change the morpho-functional characteristics of the artery wall. For example, Kawasaki disease (KD) is a vasculitis of medium- and small-caliber vessels affecting the preschool child, whose most fearsome complication is coronary aneurysms, with the possibility of partial or total secondary obstruction. It can also be associated with myocardial infarction and ischemic heart disease, and, more generally, patients are exposed to increased CV morbidity. Alterations in the structure and function of the arterial wall are also observed in adults born preterm, in children with congenital heart disease, or undergoing chemo-radiotherapy treatment for neoplasia, and even subjects with systemic diseases, such as systemic lupus erythematosus. A picture of multisystem inflammation with major cardiovascular involvement, Multisystem Inflammatory Syndrome in Children (MIS-C), is a rare but potentially fatal complication of SARS-CoV-2 infection in children, in which endothelial damage plays a central pathogenetic role and its possible association with arterial stiffness has been postulated, but studies on it are few. Detecting increased arterial stiffness as early as in children and adolescents could have important clinical repercussions for the above.

On the one hand, it would make it possible to stratify patients according to CV risk, also with a view to personalized medicine. It could allow the identification of new associations between certain diseases or exposure to environmental factors and increased arterial stiffness. Finally, it would allow assessment of the effectiveness of therapies: treatment from the earliest stages of functional impairment could change the natural history of disease, and consequently CV morbidity and mortality at later ages. VICORDER© is a quick and easy-to-use oscillometric device for studying vascular function by measuring, among other parameters, PWV. Its use in noninvasive measurement of PWV has been studied and validated in both adults and children and adolescents. In particular, the validation study by Kracht et al. was conducted in 156 children between 6 and 18 years of age, with the finding of excellent intra- and inter-observer repeatability, ease of use and tolerability for patients, making it suitable for large-scale studies. The study by Thurn et al. was conducted on 1003 healthy patients between 6 and 18 years of age and established normal PWV values (by sex, age, and height) measured with VICORDER© in pediatric age.

The device takes the form of a series of cuffs, similar in every way to a traditional sphygmomanometer, connected to a computer for analysis. The test involves the serial inflation and deflation of these cuffs, using an automatic procedure similar to that of measuring blood pressure with a digital sphygmomanometer.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 6 to 17 years of age (extremes included) being treated in the Outpatient Departments of Emergency Pediatrics or admitted to the Department of Emergency Pediatrics
* Patient cooperation during the performance of the examination.
* Obtaining informed consent from the parent/legal guardian

Exclusion Criteria:

* Behavioral disorders or severe cognitive retardation, extreme agitation, or other factors that may impair the proper performance of the examination.
* Anatomical alterations or presence of device or local pathology that conflicts with the placement of the VICORDER© cuffs.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Vascular properties, and in particular arterial stiffness, will be studied in control patients or patients with cardiovascular risk factors and comorbidities, aged 6 to 17 years (extremes included).
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06-18 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Check whether pediatric patients with CV risk factors have increased arterial stiffness compared with patients without risk factors. | through study completion, an average of 1 year
  Check whether pediatric patients with CV risk factors have increased arterial stiffness compared with patients without risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Fabi, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero - Universitaria di Bologna, U.O. Pediatria d'Urgenza, Pronto Soccorso e Osservazione Breve ed Intensiva, Bologna, Italy